CLINICAL TRIAL: NCT00850681
Title: A Randomized, Controlled Study to Evaluate the Photoallergic Potential of PEP005 (Ingenol Mebutate) Gel, 0.01% in Healthy Volunteers Using an Open Application Photoallergic Test Design
Brief Title: A Study to Evaluate the Photoallergic Potential of PEP005 (Ingenol Mebutate) Gel, 0.01% in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peplin (Industry)
Responsible Party: Robert Whitfield, Peplin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEP005-024
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2009-04

CONDITIONS: Actinic Keratosis
Keywords: Peplin; PEP005
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): PEP005 (ingenol mebutate) Gel
  Interventions: Drug: PEP005 (ingenol mebutate) Gel

INTERVENTIONS:
Drug: PEP005 (ingenol mebutate) Gel — PEP005 (ingenol mebutate) Gel, 0.01%

SUMMARY:
This Phase 1 study is designed to determine the photoallergic potential of PEP005 Gel, 0.01% and it's vehicle on normal skin.

ELIGIBILITY:
Inclusion Criteria:

* are healthy males or females;
* in the case of females of childbearing potential, are using an acceptable form of birth control and provide a negative urine pregnancy test;
* read, understand and provide signed informed consent.

Exclusion Criteria:

* are not willing to refrain from using topical/systemic analgesics within 72 hours prior to and during the study;
* are using systemic/locally-acting medications during the study and within 2 weeks prior to the beginning of the study;
* are using systemic/locally-acting anti-inflammatories during the study and within 72 hours prior to the beginning of the study;
* have participated in any clinical testing of an investigational drug within 28 days or any clinical patch application within 14 days prior to enrollment or are currently participating in any clinical testing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To determine the photoallergic (sensitizing) potential of PEP005 Gel and it's vehicle on normal skin. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jonothan S Dosik, MD, Principal Investigator — TKL Research, Inc.
Locations (1):
- TKL Research, Inc., Paramus, New Jersey, United States

REFERENCES:
- [Derived] Dosik JS, Damstra M, Udell C, Welburn P. Evaluation of the skin sensitization, photoirritation, and photoallergic potential of ingenol mebutate gel in healthy volunteers. J Clin Aesthet Dermatol. 2014 Apr;7(4):35-42. PMID 24765228
- See also: Food and Drug Authority — http://www.fda.gov